CLINICAL TRIAL: NCT06438328
Title: Effectiveness of Scapular Muscle Training in Improving Grip Strength Among Lateral Epicondylitis Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Muhammad Naveed Babur (Other)
Responsible Party: Sponsor-Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Organization: Superior University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MSRSW/Batch-Fall22/710
Record Dates: First submitted 2024-05-20; First posted 2024-05-31 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Lateral Epicondylitis
MeSH Terms: conditions — Tennis Elbow | interventions — Hand Strength

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Left/ Right affected arm (Active Comparator)
  Interventions: Diagnostic Test: Left/ Right affected arm
- Grip strength (Other)
  Interventions: Other: Grip strength

INTERVENTIONS:
Diagnostic Test: Left/ Right affected arm — Therapeutic exercises: eccentric and concentric exercises and wrist isometrics 10 repetitions of 3 sets with 10 seconds interval
  Arms: Left/ Right affected arm
Other: Grip strength — assessed by using modified sphygmomanometer in which it first inflated to 100 mmHg with closed valve. The pressure was reduced to 20mmHg and the resisted wrist extension performed at baseline and at the 4th week.
  Arms: Grip strength

SUMMARY:
The effectiveness of scapular muscular training along with conventional physiotherapy on the improving the grip strength of the patients suffering with the lateral epicondylitis was assessed by diving 56 patinets in two grousp as Group A (n=28) was treated with conventional physiotherapy treatment and Group B (n=28) was treated with Scapular strengthening and conventional physiotherapy protocol.

ELIGIBILITY:
Inclusion Criteria:

* Age: 20-50 years
* Gender: Male and Female
* Pain on the lateral epicondyle
* VAS scoring more than 4
* Positive test: Tomson test, Mill's test , Cozen;s sign and Maudsley's test

Exclusion Criteria:

* Any neurological/ Radiculopathy signs in upper limb
* Cervical pain
* Bilateral elbow pain
* History of elbow or wrist surgery
* Receiving any corticosteroid injection within last 6 months

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Severity of Disability | 12 Months
  Measured by Patient-Rated Tennis Elbow Evaluation (PRTEE)from the scoring between 0-100 at baseline and at the 4th week.
Grip strength: | 12 months
  assessed by using modified sphygmomanometer in which it first inflated to 100 mmHg with closed valve. The pressure was reduced to 20mmHg and the resisted wrist extension performed at baseline and at the 4th week.

CONTACTS AND LOCATIONS:
Locations (1):
- Fatima medical center near green town, Bhakkar, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No